CLINICAL TRIAL: NCT05390463
Title: Feasibility of the PERformance Guided Fracture Rehablitation Method (PERFoRM) Protocol for Periarticular Upper Extremity Fractures
Brief Title: Feasibility of the PERformance Guided Fracture Rehablitation Method-protocol
Acronym: PERFoRM
Status: Completed | Type: Observational
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: Z2021143
Record Dates: First submitted 2022-03-22; First posted 2022-05-25 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Fracture of Proximal End of Humerus; Fracture of Distal End of Radius; Upper Extremity Fracture; Upper Limb Fracture
Keywords: Fracture; Upper extremity; Radius; Humerus; Surgery; Rehabilitation; Surgical fixation; Protocol
MeSH Terms: conditions — Fractures, Bone | interventions — Clinical Protocols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PERFoRM: Patients with surgically treated peri-articular fractures of the upper extremity (proximal humerus and distal radius fractures) undergoing treatment within the MDTU (Multi Disciplinary Trauma Unit) of the Zuyderland MC in Heerlen are included in this study.
  Interventions: Other: PERformance guided Fracture Rehablitation Method (PERFoRM) protocol.

INTERVENTIONS:
Other: PERformance guided Fracture Rehablitation Method (PERFoRM) protocol. — A structured rehabilitation protocol for surgically treated peri-articular fractures of the upper extremity (proximal humerus and distal radius fractures).

SUMMARY:
Introduction: The scientific support for prescribed rehabilitation programs for upper extremity fractures is scarce, early mobilization has previously been shown to benefit the speed of recovery at the activity and participation level. Different (inter)national protocols for fracture rehabilitation of the upper extremity are not very specific with regard to the content of (para)medical treatment. The above underlines the need for a clearly defined and practically feasible treatment method.

That is why the PERformance guided Fracture Rehablitation Method (PERForRM) protocol was drawn up, in which the treatment method is clearly described in a structured and protocol-based manner. The ultimate goal of the PERformance guided Fracture Rehablitation Method (PERFoRM) protocol is to optimize recovery, with maximum recovery of activity and participation level in upper extremity fractures. Expert opinion/empiricism was used during the writing of the protocol, partly arising from the earlier development of a protocol for the lower extremity. The approach according to the PERForRM protocol does not focus on the time-contingent load on the fracture, but rather on the functional use of the extremity, whereby the quality of movement is paramount. The PERForRM protocol proposes a "gold standard" in the form of milestones for describing the quality of movement of the upper extremity for (para)medics.

Method:

The aim of this pilot study is to test the manageability/feasibility of this protocol in clinical practice in patients with peri-articular fractures of the upper extremity (proximal humeral and distal radius fractures). It also describes the recovery in the area of the ICF domains and the complications that occurred when applying the PERForRM protocol. The inclusion period consists of 3 months, with a follow-up of 6 months. The manageability is measured by means of a questionnaire that is administered to the practitioners (2x during the study period). The data analysis will mainly have a descriptive character

DETAILED DESCRIPTION:
Research question:

Question 1: How has the feasibility of the PERFORM protocol been applied in patients with peri-articular fractures of the upper extremity (operated proximal humeral and distal radius fractures)? Question 2a: How is the recovery on the different ICF domains after applying the PERFORM protocol in patients with peri-articular fractures of the upper extremity (proximal humeral and distal radius fractures) compared to results already described in the literature with regard to recovery (semi-structured treatment / protocols) after related fractures? Question 2b: Is the number of complications occurring when applying the PERFORM protocol equal to the results already described in the literature with regard to recovery (semi-structured treatment / protocols) after the relevant fractures?

Hypothesis:

Question 1: The PERForRM protocol can be used by both physicians and paramedics in the trauma rehabilitation chain. Experiences of physicians and paramedics show that the protocol is useful and applicable within the patient population (patients with peri-articular fractures of the upper extremity (operated proximal humeral and distal radius fractures)).

Question 2a: Patients with peri-articular fractures of the upper extremity treated with the PERFORM protocol show comparable or faster recovery in the different ICF domains compared to patients with peri-articular fractures of the upper extremity (proximal humerus). - and distal radius fractures) treated with a different post-treatment protocol (often diverse and semi- or only globally structured) as described in the literature.

Question 2b: A comparable number of complications occur in the study population and recovery in the different ICF domains is as fast or faster compared to results from the literature already described (Quick-DASH, JAMAR, NPRS, RAND-36).

Goal:

The aim of this study is to gain insight into the feasibility of the PERFORM protocol in patients with peri-articular fractures of the upper extremity (operated proximal humeral and distal radius fractures). The patients receive care-as-usual, but structured and recorded according to the PERForRM protocol. In addition, the aim of this study is to document the recovery of the patient population at the ICF level with a structured follow-up treatment according to the PERFORM protocol.

Method:

The manageability of the PERForRM protocol is investigated in a prospective, observational study design. Patients with upper extremity fractures are included post-operatively and treated according to the PERFORM protocol for 3 months. Measurement moments are 0-2, 6, 12 weeks and 6 months after the fracture. The paramedical treatment will last 3 months, after which, depending on the performance level at that time, an advice will be issued regarding aftercare.

The inclusion will take place within the MDTU (MultiDisciplinary Trauma Unit) of the Zuyderland MC in Heerlen by the specialties surgery and orthopedics and the associated (trauma) surgeons and orthopaedists. The application of the paramedical treatment will take place within the Rehabilitation Department of the Zuyderland MC at the Heerlen location.

Study population:

Patients with operated peri-articular fractures of the upper extremity (proximal humerus and distal radius fractures) who are undergoing treatment within the MDTU (Multi Disciplinary Trauma Unit) of the Zuyderland MC in Heerlen are included in this study.

Number of intended subjects:

Given the limited number of intended subjects and the heterogeneity of the group and the lack of a normal distribution of the descriptive prospective pilot study, a sample size calculation is not realistic. In view of the feasibility of the pilot study within the Rehabilitation Department, an estimate was made with regard to the inclusion number of a maximum of 30 subjects. The maximum number of 30 subjects was chosen because of the practical feasibility and treatment capacity of the rehabilitation outpatient clinic.

Data collection:

Research question 1: Two qualitative measurements were performed to test the practicality of the PERForRM protocol. The feasibility of the PERForRM protocol is recorded twice via a standardized questionnaire with the practitioner (start and end of the pilot).

Research question 2 (2a/2b): PAG = pt ass guide; AIG = aims ident guide; TEG = treatment evaluation guide; Milestones = standardized list of skills to be achieved; (quick-)DASH = disab arm should hand; JAMAR = JAMAR hand dynamometer; NPRS = num pain rating scale; RAND-36 = research and develop-36; general health condition.

Collecting data:

The medical information is collected by the doctors involved in this study The paramedical information is collected by the paramedics involved.

Data Inspection:

Given the predominantly descriptive nature of this pilot study and the existing experience with treatment as described in the protocol, no extreme qualitative or quantitative values are expected. If this is the case, the pilot should be able to detect these kinds of effects. If missing values arise in the questionnaires, reminders are sent repeatedly to encourage people to provide missing data.

Testing for normal distribution:

Since this study is a pilot study, as a result of which the number of participants is so low and the patients with their fractures are so heterogeneous, it is expected that the data will not be distributed according to a normal distribution. This is tested by means of the Shapiro-Wilk test.

Descriptive statistics:

For the normally distributed data, the mean +/-SD will be reported and students' t-test will be used for comparisons. For non-parametric data, we will report the median +/- interquartile range (IQR) and use the Mann Whitney U tests. The descriptive statistics of the results of the survey data are presented in tables. From there, the ordinal values will be used to calculate means, median, and dispersion. The nominal values will be shown in percentages of the whole.

(Interim) analyses: After completion of the rehabilitation, the data is processed and further descriptive. At the end of the 3-month follow-up, data are completed and added anonymously to the complete data set. Given the predominantly descriptive nature of the study, we do not expect extensive analyses, this will be limited to: Discriptives, T-Test (comparison T0, T1, T2, T3).

Coding and Interpreting:

The experiences of the (para)medics will be collected in the form of a questionnaire. The research group collects these experiences, which are then displayed anonymously. Subsequently, the qualitative data is coded and categorized and interpreted by means of a code tree.

Software:

Software that is used for registering data is data manager and for analyzing the results Excel and/or SPSS.

Data management:

* Location: the research data is initially collected in the patient file. From the patient file, this data is extracted to data manager and, if necessary, exported to Excel/SPSS.
* Retention of data: The data associated with this study will be kept for 15 years.
* Security of data: the research data as stated in the patient file are only accessible to the (para)medics involved. Data-manager is accessible to all members of the research team.
* Coding: the coding takes place after the patient has completed the informed consent. Numbers from 1 to 100 are assigned to the patient's hospital identification number and are saved in a new Excel file. This will be done for one of the researchers.
* Code key: The code key is stored on a server at Medisch Centrum Zuyderland. Only listed researchers have access to the code key.

Protection of privacy

* The privacy of the participants is protected from the basic agreements for the use of the patient file. Furthermore, no data is recorded in places other than the patient file or data manager.
* Sharing data: The data is not shared with institutions or persons outside Zuyderland. Results of the pilot in general, in the form of a scientific presentation/publication, are shared with institutions/persons outside Zuyderland. However, these are not micro-level data, but macro-level data that provide answers to the research questions.

ELIGIBILITY:
Inclusion and exclusion criteria:

The inclusion criteria:

* Patients with a surgically treated (osteosynthesis) proximal humeral or distal radius fracture
* Patients aged 18 to 70 years
* Patients with a premorbid level with at least independent living and independence in ADL and/or HDL.
* Patients are able to come to the Rehabilitation outpatient clinic of the Zuyderland MC in Heerlen for treatment
* Patients are sufficiently instructable with regard to communication/language (NL/English)

The exclusion criteria:

* Multiple fractures to 1 limb
* Pathological fractures
* Complications such as trophic dysregulation/CRPS at the time of inclusion
* Extensive concomitant neurovascular injury at the time of inclusion
* Cognitive problems with regard to learnability and instructability
* Influencing psychological problems or active substance use (with the exception of injury/trauma-related (movement) anxiety, event PTSD)
* Influencing other problems/comorbidities to upper extremity such as neuromuscular disorders and anatomic anomalies
* The subject is not prepared to conform to the informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population:
  Patients with surgically treated peri-articular fractures of the upper extremity (proximal humerus and distal radius fractures) treated within the MDTU (Multi Disciplinary Trauma Unit) of the Zuyderland MC in Heerlen are included in this study.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-04-24 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of the PERFoRM-protocol at starting point of the study: qualitative assessment through standardized questionnaire. | at starting point of the study (before the first inclusion); at 0 months.
  Feasibility of the PERFoRM-protocol: qualitative assessment through standardized questionnaire (questionnaire composed by investigator).
Feasibility of the PERFoRM-protocol at 6 months after the starting point of the study: qualitative assessment through standardized questionnaire. | 6 months after above-mentioned starting point of the study.
  Feasibility of the PERFoRM-protocol: qualitative assessment through standardized questionnaire (questionnaire composed by investigator).

SECONDARY OUTCOMES:
Change of rate of disability of (affected) arm-shoulder-hand. | Change between immediate phase (0-2 weeks) post-surgery, 6 weeks post-surgery, 3 months post-surgery, 6 months post surgery.
  Measurement of change in rate of disability of (affected) arm-shoulder-hand, through (Quick-) DASH; Disability Arm Shoulder Hand - questionnaire.
  Scoring: range 0-100. Score 0: no limitations in functioning. Score 100: high limitations in functioning.
Change in handstrength of affected limb. | Change between immediate phase (0-2 weeks) post-surgery, 6 weeks post-surgery, 3 months post-surgery, 6 months post surgery.
  Measurement of change in handstrength of affected limb, through hand-held-dynamometer.
  Reference table handstrength:
  * Men: 0kg (lowest strength) - 64kg (highest strength);
  * Women: 0kg (lowest strength) - 39kg (highest strength).
Change in pain of affected limb. | Change between immediate phase (0-2 weeks) post-surgery, 6 weeks post-surgery, 3 months post-surgery, 6 months post surgery.
  Measurement of change in pain of affected limb, through Numeric Pain Rating Scale (NPRS).
  Scoring: range 0-10. Score 0: no pain. Score 10: worst pain ever.
Change in general health status. | Change between immediate phase (0-2 weeks) post-surgery, 3 months post-surgery, 6 months post surgery.
  Measurement of change in general health status, through Research and develop-36; general health status (RAND-36) - questionnaire.
  Scoring: range 0-100. Higher scores present better general health status.

CONTACTS AND LOCATIONS:
Overall Officials: MPM Dremmen, MD, Principal Investigator — Zuyderland Medisch Centrum
Locations (1):
- Zuyderland Medisch Centrum, Heerlen, Netherlands

IPD SHARING:
Plan to Share IPD: No